CLINICAL TRIAL: NCT07063628
Title: Comparative Assessment of Triglyceride-Glucose Indices and Left Ventricular Speckle Tracking in Predicting Coronary Artery Disease Severity: Insights From Gensini Scoring
Brief Title: Triglyceride-Glucose Indices and Left Ventricular Speckle Tracking in Predicting Coronary Artery Disease Severity
Status: Completed | Type: Observational
Sponsor: Damanhour University (Other)
Collaborators: Tanta University (Other)
Responsible Party: Principal Investigator, Rehab Werida, Associate Professor, Damanhour University
Other Study IDs: Predicting CAD Severity
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: TyG-derived index. — Derived indices included:
  * Ty,G×B,M,I = TyG index × body mass index
  * TyG×W,C = TyG index × waist circumference
  * TyG×WH,tR = TyG index × waist-to-height ratio Quartile-based stratification was applied to each TyG-derived index.
  Other Names: TG index
Diagnostic Test: Left Ventricular Speckle Tracking — Coronary Angiography and Gensini Scoring: All participants underwent standard diagnostic coronary angiography. CAD was categorized as one-, two-, or three-vessel disease based on the number of vessels with ≥50% stenosis. The severity of CAD was quantified using the Gensini score, which assigns a severity weight to each lesion depending on degree of stenosis and anatomical location. Final scores were calculated by summing weighted values across all coronary segments.
  Other Names: Echocardiographic Assessment

SUMMARY:
Our study specifically will address the value of modified triglyceride glucose indices versus left ventricular speckle tracking in prediction of severity of coronary artery disease assessed by Gensini score.

DETAILED DESCRIPTION:
A cross sectional study that will be conducted in Cardiovascular Department of Tanta University in Egypt in the period from May to July 2025 . Two hundred patients diagnosed with coronary artery diseases were included in the study. Patients were considered to have confirmed coronary artery disease through angiographically proven CAD.

Provision of privacy:

Privacy of all data is guaranteed and there will be a code number for every patient and include all of his or her investigations.

Informed consent:

Informed written consent will be obtained from all patients after full explanation of benefits and risks of the study.

Methods: Study patients and procedures:

Selection criteria included any patient with chronic stable angina and proved coronary artery disease by coronary angiography Exclusion criteria included: Any patients with acute coronary syndrome, arrhythmias, previous Percutaneous coronary intervention (PCI) or Coronary Artery Bypass Graft (CABG) surgery

All the participants were subjected to following:

1. History taking for presence of risk factors of cardio vascular disease as age, sex, smoking, physical inactivity, diabetes and hypertension.
2. Physical examination including height, weight and waste circumference
3. Resing 12 leads ECG
4. Laboratory investigations:

   * Fasting blood glucose (FBG)
   * Triglyceride (TG), TG index.
   * Total Cholesterol level
   * Renal Function test . Echocardiographic evaluation

6. Coronary angiography 7. Gensini score calculated by summation of the individual coronary segment scores.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of CAD with ≥50% stenosis in at least one major coronary artery.

Exclusion Criteria:

* Patients with acute coronary syndrome, arrhythmias, previous coronary interventions (PCI or CABG), or inability to undergo echocardiographic assessment.

Ages: 38 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Two hundred adult patients with chronic stable angina and angiographically confirmed coronary artery disease (CAD) were enrolled.
Sampling Method: Probability Sample
Enrollment: 508 (Actual)
Dates: Start 2025-04-30 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-03 (Actual)

PRIMARY OUTCOMES:
triglyceride-glucose (TyG) index | 2 months
  predictive value of the triglyceride-glucose (TyG) index and its modified forms (TyG×BMI, TyG×WC, TyG, ×, W,Ht,R ) with global longitudinal strain (GLS) in assessing coronary artery disease (CAD) severity, as quantified by the Gensini score.
longitudinal strain (GLS) | 2 months
  Echocardiography parameter in assessing coronary artery disease (CAD) severity
Gensini score. | 2 months
  Score assessing coronary artery disease (CAD) severity

CONTACTS AND LOCATIONS:
Overall Officials: Eman Elshaikh, Ass. Prof., Principal Investigator — Tanta University
Locations (1):
- Rehab Hussein Werida, Damanhūr, Elbehairah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siverio-Morales O, Mora-Fernandez C, Hernandez-Carballo C, Martin-Nunez E, Gonzalez-Luis A, Martin-Olivera A, Navarro-Gonzalez JF, Donate-Correa J. Predictive value of triglyceride-glucose index for the evaluation of coronary artery disease severity and occurrence of major adverse cardiovascular events. Am J Physiol Heart Circ Physiol. 2025 Jan 1;328(1):H14-H20. doi: 10.1152/ajpheart.00684.2024. Epub 2024 Nov 19. PMID 39560964
- [Background] Lopez-Jaramillo P, Gomez-Arbelaez D, Martinez-Bello D, Abat MEM, Alhabib KF, Avezum A, Barbarash O, Chifamba J, Diaz ML, Gulec S, Ismail N, Iqbal R, Kelishadi R, Khatib R, Lanas F, Levitt NS, Li Y, Mohan V, Mony PK, Poirier P, Rosengren A, Soman B, Wang C, Wang Y, Yeates K, Yusuf R, Yusufali A, Zatonska K, Rangarajan S, Yusuf S. Association of the triglyceride glucose index as a measure of insulin resistance with mortality and cardiovascular disease in populations from five continents (PURE study): a prospective cohort study. Lancet Healthy Longev. 2023 Jan;4(1):e23-e33. doi: 10.1016/S2666-7568(22)00247-1. Epub 2022 Dec 12. PMID 36521498
- [Background] Zhao S, Yu S, Chi C, Fan X, Tang J, Ji H, Teliewubai J, Zhang Y, Xu Y. Association between macro- and microvascular damage and the triglyceride glucose index in community-dwelling elderly individuals: the Northern Shanghai Study. Cardiovasc Diabetol. 2019 Jul 25;18(1):95. doi: 10.1186/s12933-019-0898-x. PMID 31345238